CLINICAL TRIAL: NCT03343444
Title: Safety & Efficacy of Sofosbuvir 400mg/Ledipasvir 90mg in the Treatment of Chronic Hepatitis C Adolescents
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED-ELH-2017
Record Dates: First submitted 2017-03-27; First posted 2017-11-17 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; ledipasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Active Comparator): Treatment-naïve is defined as having never received treatment for HCV with any interferon (IFN), ribavirin , or other approved or experimental HCV specific direct acting antivirals.
  Interventions: Drug: 12 weeks (Sofosbuvir 400mg/Ledipasvir 90mg)
- Arm 2 (Active Comparator): Treatment-experienced is defined as:
  1. IFN Intolerant
  2. Non-response
  3. Relapse/Breakthrough
  Interventions: Drug: 12 weeks (Sofosbuvir 400mg/Ledipasvir 90mg)
- Short Track (Experimental): Treatment-naïve or Treatment-experienced who achived very rapid virological responce - Negative HCV PCR after treatment with (Sofosbuvir 400mg/Ledipasvir 90mg) for 1 week
  Interventions: Drug: 8 weeks (Sofosbuvir 400mg/Ledipasvir 90mg)

INTERVENTIONS:
Drug: 12 weeks (Sofosbuvir 400mg/Ledipasvir 90mg) — Single Tablet (Sofosbuvir 400mg/Ledipasvir 90mg) daily for 12 weeks
  Other Names: Normal track
  Arms: Arm 1; Arm 2
Drug: 8 weeks (Sofosbuvir 400mg/Ledipasvir 90mg) — Single Tablet (Sofosbuvir 400mg/Ledipasvir 90mg) daily for 8 weeks
  Other Names: Short track
  Arms: Short Track

SUMMARY:
Randomized, open-label study in treatment naïve and treatment experienced, adolescence to determine the efficacy of Sofosbuvir 400mg/ledipasvir 90mg in treatment naïve and treatment-experienced adolescence. Hepatitis C virus (HCV) infection as measured by the proportion of subjects with sustained viral response 12 weeks after discontinuation of therapy (SVR12)

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. 12-18 years
3. HCV RNA ≥ 104 IU/mL at screening.
4. Confirmed chronic HCV infection as documented by either:

   a. a positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or
5. Screening ECG without clinically significant abnormalities.
6. Patients must have the following laboratory parameters at screening:

   * ALT (Alanine transaminase) ≤ 10 x the upper limit of normal (ULN)
   * AST (Aspartate Aminotransferase) ≤ 10 x ULN
   * Hemoglobin ≥ 12 g/dL for male, ≥ 11 g/dL for female patients
   * Platelets > 50,000 cells/mm3
   * INR (international normalized ratio) ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * Albumin ≥ 3 g/dL
   * HbA1c ≤ 10%
   * Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation
7. Patient has not been treated with any investigational drug or device within 30 days of the screening visit.

Exclusion Criteria:

1. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis).
2. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
3. History of solid organ transplantation.
4. Current or prior history of clinical hepatic decompensation (eg, ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome and hepatopulmonary syndrome).
5. History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
6. History of a gastrointestinal disorder (or post-operative condition) that could interfere with the absorption of the study drug.
7. History of significant pulmonary disease, significant cardiac disease or porphyria.
8. History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
9. Donation or loss of more than 400 mL blood within 2 months prior to Baseline/Day 1.
10. Known hypersensitivity to the study investigational medicinal product, the metabolites, or formulation excipients.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 12 weeks after discontinuation of therapy
  sustained viral response 12 weeks after discontinuation of therapy (SVR12)

SECONDARY OUTCOMES:
SVR4 | 4 weeks after discontinuation of therapy
  sustained viral response 4 weeks after discontinuation of therapy (SVR4)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Shiha, MD, Principal Investigator — Egyptian Liver Hospital
Locations (1):
- Egyptian Liver Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No